CLINICAL TRIAL: NCT02946424
Title: Simvastatin to Improve Bone Health in SCI: A Double-Blind, Randomized, Placebo-Controlled Clinical Trial
Brief Title: Simvastatin to Prevent SCI-Induced Bone Loss
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Craig Hospital (Other)
Responsible Party: Principal Investigator, Leslie Morse, Principal Investigator, Craig Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SCIMS Statin
Record Dates: First submitted 2016-10-13; First posted 2016-10-27 (Estimated); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Spinal Cord Injuries; Osteoporosis
MeSH Terms: conditions — Spinal Cord Injuries; Osteoporosis | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Simvastatin treatment (Experimental): Simvastatin for one year time period
  Interventions: Drug: Simvastatin
- Placebo treatment (Placebo Comparator): Placebo for one year time period
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Placebo Oral Capsule — 12 month course of daily placebo
  Arms: Placebo treatment
Drug: Simvastatin — 12 month course of daily simvastatin
  Other Names: Zocor
  Arms: Simvastatin treatment

SUMMARY:
This is a double blind, randomized, placebo -controlled clinical trial with the primary goal of determining the osteogenic benefits of simvastatin in acute SCI.

DETAILED DESCRIPTION:
Investigators will test if a 1- year course of simvastatin (40 mg daily) will prevent bone loss compared to placebo in the first year following SCI.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age
* acute SCI (AIS A-C) who are enrolled at our center in an ongoing surveillance study.
* use a wheelchair as their primary mobility mode
* reside in the greater Denver metropolitan area
* within 3 months of injury
* medically stable
* able to follow directions
* provide informed consent.

Exclusion Criteria:

- have any simvastatin contraindications including:

* drug allergy,
* active liver disease,
* renal dysfunction,
* concurrent use of drugs that cause myopathy or increase the risk of myopathy with simvastatin therapy (gemfibrozil, niacin, cyclosporine, danazol, amiodarone, dronedarone, ranolazine, calcium channel blockers, colchicine), strong CYP34A inhibitors (itraconazole, ketoconazole, posaconazole, voriconazole, erythromycin, clarithromycin, telithromycin, HIV protease inhibitors, boceprevir, telaprevir, nefazodone, cobicistat-containing products), low plasma cholesterol levels,
* uncontrolled or poorly controlled diabetes,
* unstable anti-coagulation treatment,
* taking a statin in the preceding 12 months,
* metabolic bone disease, thyroid disorder,
* history of bilateral oophorectomy,
* current use of medications potentially affecting bone health including bisphosphonates, androgenic steroids, estrogenic steroids, anti-epileptics, lithium glucocorticoid use for more than 3 months,
* have received inhaled glucocorticoids in the past 12 months,
* pregnant or lactating women,
* women of childbearing potential who are unwilling or unable to use a reliable form of contraception.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in knee bone mineral density | baseline and 12 months
  assessed by DXA

SECONDARY OUTCOMES:
Change in bone volume | baseline and 12 months
  quantitative CT scan of the knee
Change in mood | baseline and 12 months
  Patient Health Questionnaire-9
Change in pain | baseline and 12 months
  International Spinal Cord Injury Basic Pain Data Set
Satisfaction with life | baseline and 12 months
  Satisfaction with Life Scale
Change in community reintegration | baseline and 12 months
  Craig Handicap and Assessment Reporting Technique-Short Form
Change in motor score | baseline and 12 months
  assessed by ISNCSCI exam
Change in tibial bone strength | baseline and 12 months
  assessed by finite element analysis of quantitative CT scan of the knee

OTHER OUTCOMES:
Change in bone formation | baseline and 12 months
  assessed by circulating osteocalcin level
Change in bone resorption | baseline and 12 months
  assessed by circulating c-telopeptide level

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Morse, DO, Principal Investigator — Craig Hospital
Locations (1):
- Craig Hospital, Englewood, Colorado, United States

REFERENCES:
- [Derived] Kowalski JL, Nguyen N, Battaglino RA, Falci SP, Charlifue S, Morse LR. miR-338-5p Levels and Cigarette Smoking are Associated With Neuropathic Pain Severity in Individuals With Spinal Cord Injury: Preliminary Findings From a Genome-Wide microRNA Expression Profiling Screen. Arch Phys Med Rehabil. 2022 Apr;103(4):738-746. doi: 10.1016/j.apmr.2021.09.005. Epub 2021 Oct 27. PMID 34717922